CLINICAL TRIAL: NCT01854437
Title: The Effect of Magnesium Oxide on Plasma Phosphate in Hemodialysis Patients
Status: Completed | Type: Observational
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Maryam Pakfetrat, associated professor of shiraz Shiraz University of Medical Sciences, Shiraz University of Medical Sciences
Other Study IDs: 1391
Record Dates: First submitted 2013-05-04; First posted 2013-05-15 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2013-05

CONDITIONS: Hyperphosphatemia
Keywords: mg oxide; hyperphosphatemia; plasma phosphor level
MeSH Terms: conditions — Hyperphosphatemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Mg Oxide: Mg Oxide (Mg®, 21st Century®) 250 mg orally for 4 weeks
  Interventions: Drug: Mg Oxide
- placebo: placebo 1 tab TDS

INTERVENTIONS:
Drug: Mg Oxide — 250 mg orally for 4 weeks
  Other Names: (Mg®, 21st Century®)
  Groups: Mg Oxide

SUMMARY:
Hyperphosphatemia is a common problem in hemodialysis (HD) patients. Different chelators for control of Hyperphosphatemia are used. The aim of this study was to assess the effect of magnesium oxide (Mg Oxide) on the control of serum phosphorus (P) level and evaluation of its side effects in hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

hemodialysis with duration>3 months serum P level >5.5 mg/dl serum Ca>8 mg/dl.

Exclusion Criteria:

Mg level >3 mg/dl

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: hemodialysis patients
Sampling Method: Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2012-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
plasma phosphate level | 4 week

CONTACTS AND LOCATIONS:
Locations (1):
- Shiraz University Hemodialysis Center, Shiraz, Fars, Iran